CLINICAL TRIAL: NCT01380288
Title: Changes of Cognitive Function in Patients With Mild to Moderate Alzheimer's Disease Associated With or Without White Matter Changes After Rivastigmine Patch Therapy - Multi-center, Prospective, Open-label Clinical Trial
Brief Title: Cognitive Changes in Alzheimer's Disease Patients Associated With or Without White Matter Changes After Rivastigmine
Acronym: CAREER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dong-A University (Other)
Collaborators: Novartis Korea Ltd. (Industry)
Responsible Party: Principal Investigator, Kyungil Park, Assistant professor, Dong-A University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: neuropark
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; rivastigmine patch; white matter change
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- without white matter change (Active Comparator)
  Interventions: Drug: rivastigmine patch
- with white matter change group (Active Comparator)
  Interventions: Drug: rivastigmine patch

INTERVENTIONS:
Drug: rivastigmine patch — rivastigmine patch 5cm2 for 4 weeks and then augmented to 10cm2 for 20 weeks
  Other Names: Exelon patch

SUMMARY:
The purpose of this study is to evaluate and compare the changes of cognitive function (as measured by ADAS-Cog) in the two group of patients with Alzheimer's disease (AD) associated with and without white matter changes after rivastigmine patch therapy.

DETAILED DESCRIPTION:
Acetylcholinesterase inhibitors (AChEIs) increase the amount acetylcholine at ACh receptors within the brain, and are the primary medications used to treat AD. Alzheimer's disease patients are frequently associated with mild or moderate white matter changes on MR imaging. The impact of whiter matter changes on the efficacy of cognition, functional abilities, behavioral and psychiatric symptoms and caregiver burden for probable Alzheimer's disease is not well known. There are very few studies for the efficacy of rivastigmine between the patients with mild to moderate Alzheimer's disease associated with or without vascular risk factors.

Recently, the rivastigmine patch demonstrated efficacy comparable to the highest doses of rivastigmine capsules, with markedly improved tolerability profile. The investigators hypothesized that rivastigmine patch will provide benefits to AD patients with white matter changes compared to those without any white matter changes. Possible explanation about favorable benefits for AD with white matter changes is that rivastigmine may act on both Alzheimer's and vascular pathologies contributing to dementia, providing additive treatment effects in patients suffering from both conditions concurrently. To our Knowledge, there was no study or clinical trial to compare the changes of cognitive function, ADL, BPSD and caregiver burden in two groups of patient with Alzheimer's disease associated with or without white matter changes after rivastigmine transdermal patch therapy.

ELIGIBILITY:
Inclusion Criteria:

* AD in NINCDS-ADRDA criteria, mild to moderate
* probable AD with or without mild to moderate whiter matter lesions, excluding multiple large vessel infarcts or a single, strategically placed infarct (angular gyrus, thalamus, basal forebrain, territory of the posterior or anterior cerebral artery) on MRI scan (within 12 months)
* MMSE score : 10 to 26 at screening
* Hachinski scores ≤ 4
* No clinically significant laboratory abnormalities, such as thyroid disease, vitamine B12 deficiency or folic acid deficiency

Exclusion Criteria:

* Current evidence of history of neurological, psychiatric and other illness that could contribute to dementia
* Subjects with clinical significant cardiovascular disease, stroke, pulmonary disease or any other medical disease in the past 6 months
* History of cancer within the last 5 years
* Subjects with evidence or history of clinically significant allergic reaction to AchEI or drugs
* Subjects who had significant visual or hearing difficulties

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
The changes of cognitive function as measured by ADAS-Cog | 24 weeks

SECONDARY OUTCOMES:
MMSE (Mini-Mental State Examination) | 24 weeks
Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) | 24 weeks
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | 24 weeks
Caregiver-Administered Neuropsychiatric Inventory (CGA-NPI) | 24 weeks
Caregiver burden scale | 24 weeks
Adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Won Park, MD, PhD, Principal Investigator — Dong-A University
Locations (16):
- South Korea (16):
  - Holy Family Hospital, The Catholic Univerisy of Korea, School of Medicine, Bucheon-si
  - Busan National University Hospital, Busan
  - Busan Paik Hospital, Inje University College of Medicine, Busan
  - Changwon Fatima Hospital, Changwon
  - Daegu Fatima Hospital, Daegu
  - Keimyung University School of Medicine, Daegu
  - Kyungpook National University School of Medicine, Daegu
  - Myongji Hospital, Kwandong University College of Medicine, Goyang
  - Dongguk University International Hospital, Ilsan
  - National Health Insurance Corporation Ilsan Hospital, Ilsan
  - Inha University College of Medicine, Incheon
  - Gyeongsang National University College of Medicine, Jinju
  - Chonnam National University, Medical School, Kwangju
  - Seoul National Unviersity College of Medicine, Clinical neuroscience center, Seoul National Unviersity Bundang Hospital, Seongnam
  - The Catholic Univerisy of Korea, School of Medicine, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

REFERENCES:
- [Derived] Park KW, Kim EJ, Han HJ, Shim YS, Kwon JC, Ku BD, Park KH, Yi HA, Kim KK, Yang DW, Lee HW, Kang H, Kwon OD, Kim S, Lee JH, Chung EJ, Park SW, Park MY, Yoon B, Kim BC, Seo SW, Choi SH. Efficacy and tolerability of rivastigmine patch therapy in patients with mild-to-moderate Alzheimer's dementia associated with minimal and moderate ischemic white matter hyperintensities: A multicenter prospective open-label clinical trial. PLoS One. 2017 Aug 7;12(8):e0182123. doi: 10.1371/journal.pone.0182123. eCollection 2017. PMID 28786987